CLINICAL TRIAL: NCT06682156
Title: Clinical Outcome of Multiple Myeloma Patients Switching to Carfilzomib-based Regimens After Prior Bortezomib-based First-line Therapy Intolerant, a Real-world, Single-arm, Prospective Study
Brief Title: Conversion to Carfilzomib Therapy in Bortezomib Intolerant Newly Diagnosed Multiple Myeloma(NDMM) Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: Kcv-MM12
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-04

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — carfilzomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- K-based therapy: if bortezomib related intolerance happens during front line therapy of bortezomib-based triple regimen, then carfilzomib-based therapy will be used
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — carfilzomib C1: 20mg/m2，D1-2; 27mg/m2，D8-9; 36mg/m2，D15-16 C2 and subsequent cycles: 36mg/m2。
  Other Names: Kyprolis

SUMMARY:
This is an open-label, single-arm, prospective study conducted in real-world clinical practice. It aims to evaluate the efficacy and safety in Chinese patients with newly diagnosed multiple myeloma who switch to carfilzomib-based regimens after bortezomib-based triple-drug regimen intolerance happens.

DETAILED DESCRIPTION:
This is an open-label, single-arm, prospective study conducted in real-world clinical practice. Chinese patients with newly diagnosed multiple myeloma will be enrolled if they switch to carfilzomib-based regimens after bortezomib-based triple-drug regimen intolerance happens.

Induction and consolidation therapy will be 6-8cycles. 6 cycles for transplant recipients and 8 cycles for non-transplant recipients. Maintenance therapy will continue until progression.

It aims to evaluate the efficacy and safety of carfilzomib based therapy in Chinese NDMM patients with intolerance to bortezomib. The primary endpoint is the rate of 2-year pFS and secondary endpoints are the rate of ORR,sCR/CR,VGPR,PR, the rate and duration of MRD, the rate of 2-year OS and safety.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Diagnosed with multiple myeloma according to IMWG criteria.
3. Patients who have received only first-line bortezomib-based triple therapy, including bortezomib/lenalidomide/dexamethasone (VRD), bortezomib/thalidomide/dexamethasone (VTD）,bortezomib/ cyclophosphamide/dexamethasone (VCD), and bortezomib/adriamycin//dexamethasone (PAD).
4. Eastern cooperative oncology group(ECOG) score 0-2
5. Patients who develop toxicities associated with bortezomib therapy evaluated by the investigator, including the presence of Grade 1 with pain or Grade 2 peripheral neuropathy (PN), Grade 3 hepatic impairment, Grade 3 diarrhea, and any other Grade 3 non-hematologic adverse events and resulting in bortezomib dose reduction or discontinuation.
6. Patients who agree to and sign informed consents to participate in this study.

Exclusion Criteria:

1. Patients currently participating in other interventional clinical studies (except those currently participating in non-interventional observational studies)
2. Patients who have received prior carfilzomib treatment or participated in carfilzomib associated studies (with or without carfilzomib treatment).
3. Patients with a primary diagnosis of MM combined with plasma cell leukemia (peripheral blood monoclonal plasma cells ≥5% of the total number of differentiated mature leukocytes)
4. Patients who have not fully recovered from the reversible effects of prior chemotherapy (i.e., <= grade 1 toxicity).
5. Patients with other malignancies diagnosed prior to the MM diagnosis, excluding squamous and basal cell carcinomas of the skin, and carcinoma in situ of the cervix or breast, which can be cured within 3 years with minimal risk of recurrence.
6. Patients with an active systemic infection, active hepatitis B or C virus infection, or known positive test results for human immunodeficiency virus.
7. Evidence of current uncontrolled cardiovascular disease, including hypertension, arrhythmias (prolonged QT interval, ventricular tachycardia, ventricular flutter, ventricular fibrillation, frequent ventricular premature beats (24-hour premature loading of ≥15% of the total number of beats), grade Ⅲ atrioventricular block, and a heart rate of <30-40 bpm congestive heart failure, unstable angina, or myocardial infarction in the past 3 months,. New York Heart Association (NYHA) class III and IV heart failure. left ventricle ejection fraction（LVEF） <40% on cardiac ultrasound.
8. Participants with known chronic obstructive pulmonary disease (COPD) (defined as forced expiratory volume in 1 second [FEV1] <50% of predicted normal value), persistent asthma, or a history of asthma within the past 2 years (controlled intermittent asthma or mild persistent asthma that is allowed). Participants with known or suspected COPD must undergo FEV1 testing during screening.
9. Inability to comply with protocol/procedure.
10. Patients with hypersensitivity to the active ingredient or excipients of carfilzomib.
11. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed multiple myeloma patients who develop toxicities associated with bortezomib therapy evaluated by the investigator, including the presence of Grade 1 with pain or Grade 2 peripheral neuropathy (PN), Grade 3 hepatic impairment, Grade 3 diarrhea, and any other Grade 3 non-hematologic adverse events
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Outcome of peripheral neuropathy | from enrollment to 2 years
  recurrence of peripheral neuropathy

SECONDARY OUTCOMES:
ORR | from enrollment to 2 years
  the rate of sCR,CR, PR and VGPR according to IMWG（International Myeloma Working Group） criteria
sCR/CR rate | from enrollment to 2 years
  the rate of sCR/CR according to IMWG criteria
PR rate | from enrollment to 2 years
  the rate of PR according to IMWG criteria
VGPR rate | from enrollment to 2 years
  the rate of VGPR according to IMWG criteria
MRD negativity rate | from enrollment to 2 years
  the rate of minimal residual disease
AE rate | from enrollment to 2 years
  the rate of adverse events
2-year OS rate | from enrollment to 2 years
  the rate of Overall survival at 2 years
Duration of MRD negativity | from enrollment to 2 years
  Duration of minimal residual disease negativity
2-year PFS rate | from enrollment to 2 years
  the rate of progression free survival at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Lingzhi Yan, Suzhou, Jiangsu, China